CLINICAL TRIAL: NCT00784563
Title: Effects of Aerobic Exercise in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6261-R
Record Dates: First submitted 2008-10-30; First posted 2008-11-04 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Exercise/*physiology; *Physical Fitness; Rehabilitation; Cognition
MeSH Terms: conditions — Parkinson Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous training (Active Comparator): Aerobic walking using continuous heart rate training.
  Interventions: Behavioral: Continuous training
- Interval training (Active Comparator): Aerobic walking using interval heart rate training
  Interventions: Behavioral: Interval training

INTERVENTIONS:
Behavioral: Continuous training — The maximal heart rate (HRmax) in the exercise prescription was based on age[Goldberg, Elliot, and Kuehl1988] and reduced by 20% in participants who used beta-blockers.[Wonisch et al. 2003] The duration of exercise sessions (3x/week) was advanced from 15 to 45 minutes over the first 6 weeks. The goal for continuous training was to remain within 70-80% of HRmax throughout the session.
  Arms: Continuous training
Behavioral: Interval training — Interval trainees alternated every 3 minutes between slower (60-70% of HRmax) and faster (80-90% of HRmax) walking [Wisloff et al. 2007].
  Arms: Interval training

SUMMARY:
Motivated by reported improvements in aerobic fitness and executive functions after a 6-month aerobic walking intervention in normal sedentary elderly, we conducted a Phase I/II study to investigate effects of aerobic exercise on motor function, cognition, and quality of life in mild-moderate patients with Parkinson's disease (PD). To identify the best method to deliver fitness training, we also aimed to compare safety, tolerability, and fitness benefits between different training methods (continuous/moderate intensity vs. interval/alternating between low and vigorous intensity) and exercise settings (individual vs. group). Interval training reportedly facilitates higher fitness gains than continuous training. Group training may promote success through social interaction, whereas individual training offers greater flexibility.

Details of the study can be found in the publication below:

Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting.

Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG.

Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2.

PMID: 24991037

DETAILED DESCRIPTION:
Participants:

The participants were recruited in Spring 2009, 2010, and 2011 through regional newspaper advertisements and solicitations in the Movement Disorders Clinic at the University of Iowa and the Veterans Affairs Medical Center of Iowa City. We phone screened respondents and evaluated eligible candidates in-person using clinical examination, MMSE, 12-lead ECG, blood count and biochemistry, followed by graded exercise test using cycle ergometry within one week of starting the intervention. At each visit, we obtained body weight and height, heart rate and blood pressure after 5 minutes of supine rest [Goldberg et al. 1988] and after 3 minutes of standing. Throughout the study, the medications of participants continued to be managed by their treating neurologists.

Inclusion criteria: Idiopathic PD; Hoehn and Yahr Scale I-III; men or women aged 50-80; stable dopaminergic treatment regimen for at least 4 weeks prior to baseline not requiring adjustment.

Exclusion criteria: Current participation in an aerobic exercise program; Mini Mental Status Exam score <24; confounding medical, orthopedic or psychiatric disorders; cardiac abnormalities during cycle ergometry.

Design:

Initial design was a 2x2 randomized trial of different training methods (continuous vs. interval) and settings (individual vs. group). Sample size was estimated using 80% power to detect an effect size of 0.66 SD in VO2max (estimated improvement=10% /estimated SD of change=15%) within each arm at alpha=0.05 and an attrition rate of 25%.

During the first two years, the participants were randomized in blocks of four to continuous or interval training. Logistical factors (e.g., rural residence) precluded randomization to group setting, leading to convenience-based assignments in the first year, and dropping of the group setting afterwards. In the third year, all participants were assigned to the continuous arm after preliminary analyses of prior data raised safety concerns about interval training.

Intervention:

The maximal heart rate (HRmax) in the exercise prescription was based on age [Goldberg, Elliot, and Kuehl1988] and reduced by 20% in participants who used beta-blockers [Wonisch et al. 2003]. The duration of exercise sessions (3x/week) was advanced from 15 to 45 minutes over the first 6 weeks. The goal for continuous training was to remain within 70-80% of HRmax throughout the session. Interval trainees alternated every 3 minutes between slower (60-70% of HRmax) and faster (80-90% of HRmax) walking[Wisloff et al. 2007]. We emphasized that these parameters were for guidance only and that the participants should give their best effort without feeling uncomfortable or unsafe.

Participants were asked to wear electronic heart rate and walking speed monitors (Polar RS400, Kempele, Finland) and fill out diaries for each session. A trainer facilitated group training at a track and collected monitor data and exercise diaries. Trainers conducted home visits for the individual arm participants to choose walking routes (a primary outdoor route and an alternative indoor route) and orient the participant about safe exercise procedures, followed by biweekly home visits to monitor safety and compliance.

Efficacy Measures:

The participants were tested while on their usual antiparkinsonian regimen, always with adequate symptom control to allow comfortable participation in the protocol, at baseline and at the end of the intervention by evaluators blinded to the treatment arm, but not to pre-post training status.

Aerobic fitness: Oxygen uptake (VO2) was measured from expired air samples on a breath-by-breath basis during cycle ergometry. We verified maximal effort when 2 of 3 criteria were met [Balady et al. 2010]: 1) a plateau in VO2 between two or more workloads, 2) respiratory exchange ratio ≥1.10, and 3) HR > 85% of the age predicted HRmax.

Cognition: Due to sensitivity of the Eriksen's flanker task performance to changes in aerobic fitness status [Colcombe et al. 2004;Kluding et al. 2011], we chose change in Percent Increase Score (PIS) on flanker task as the primary cognitive outcome measure. Participants were asked to identify the orientation of a central arrow cue ('<' or '>'), which was flanked on both sides by two arrow cues that either pointed in the same direction (congruent: <<<<<) or a different direction (incongruent: >><>>). Using reaction times (RT) during congruent and incongruent trials, the PIS was calculated as =((RT_incongruent - RT_congruent) / RT_congruent) * 100.[Colcombe, Kramer, Erickson, Scalf, McAuley, Cohen, Webb, Jerome, Marquez, and Elavsky2004] The Stroop test was used as another measure of inhibition.

We assessed set shifting using Wisconsin Card Sorting Test and Trail-Making Test (B-A),[Uc, Rizzo, Johnson, Dastrup, Anderson, and Dawson2009] visual perception using Judgment of Line Orientation and Complex Figure Test (CFT)-Copy, verbal memory using Rey Auditory Verbal Learning Test, visual memory using CFT-Recall, language using Controlled Oral Word Association Test,[Uc, Rizzo, Johnson, Dastrup, Anderson, and Dawson2009] and general cognition using Montreal Cognitive Assessment.[Chou et al. 2010] Parkinsonism: Unified Parkinson's Disease Rating Scale and timed motor tests (7m Walk and finger tapping),[Defer et al. 1999] Functional Reach test for balance,[Uc, Rizzo, Johnson, Dastrup, Anderson, and Dawson2009] total daily levodopa equivalents,[Tomlinson et al. 2010] and a patient diary [Hauser et al. 2004].

Quality of life: Fatigue Severity Scale,[Friedman et al. 2011] Geriatric Depression Scale,[Uc, Rizzo, Johnson, Dastrup, Anderson, and Dawson2009] PD Quality of Life Scale (PDQUALIF) [Welsh et al. 2003].

Statistical analysis Two-sample t-tests, Wilcoxon Rank-Sum, or Fisher's Exact tests were used to compare baseline features and exercise characteristics and outcomes between different treatment arms, and between the completers and dropouts, and to compare baseline cognitive performance of our PD participants with controls from our driving studies.[Uc, Rizzo, Johnson, Dastrup, Anderson, and Dawson2009] Regression methods were used to adjust these comparisons for age, education, and gender.

As all treatment arms were designed to deliver a similar average aerobic intensity, we planned to pool a priori all completers throughout the study to analyze the effects of aerobic exercise with higher statistical power. We used Wilcoxon Signed Ranks tests or paired t-tests to compare final vs. baseline outcomes. When a significant change in outcomes was observed, we used regression models to assess and adjust for the effect of different settings and training methods, calendar year, and change in levodopa equivalent. We also used Pearson correlations and regression models to quantify associations of changes in outcomes with changes in aerobic fitness.

The analyses of magnetic resonance imaging studies and other biomarkers is continuing and will be published in the future.

Reference List

Balady GJ, Arena R, Sietsema K et al. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation 2010; 122: 191-225.

Chou KL, Amick MM, Brandt J et al. A recommended scale for cognitive screening in clinical trials of Parkinson's disease. Mov Disord 2010; 25: 2501-2507.

Colcombe SJ, Kramer AF, Erickson KI et al. Cardiovascular fitness, cortical plasticity, and aging. Proc Natl Acad Sci U S A 2004; 101: 3316-3321.

Defer GL, Widner H, Marie RM, Remy P, Levivier M. Core assessment program for surgical interventional therapies in Parkinson's disease (CAPSIT-PD). Mov Disord 1999; 14: 572-584.

Friedman JH, Abrantes A, Sweet LH. Fatigue in Parkinson's disease. Expert Opin Pharmacother 2011; 12: 1999-2007.

Goldberg L, Elliot DL, Kuehl KS. Assessment of exercise intensity formulas by use of ventilatory threshold. Chest 1988; 94: 95-98.

Hauser RA, Deckers F, Lehert P. Parkinson's disease home diary: Further validation and implications for clinical trials. Mov Disord 2004; 19: 1409-1413.

Kluding PM, Tseng BY, Billinger SA. Exercise and executive function in individuals with chronic stroke: a pilot study. J Neurol Phys Ther 2011; 35: 11-17.

Tomlinson CL, Stowe R, Patel S, Rick C, Gray R, Clarke CE. Systematic review of levodopa dose equivalency reporting in Parkinson's disease. Mov Disord 2010; 25: 2649-2653.

Uc EY, Rizzo M, Johnson AM, Dastrup E, Anderson SW, Dawson JD. Road Safety in Drivers with Parkinson Disease. Neurology 2009; 73: 2112-2119.

Welsh M, McDermott MP, Holloway RG, Plumb S, Pfeiffer R, Hubble J. Development and testing of the Parkinson's disease quality of life scale. Mov Disord 2003; 18: 637-645.

Wisloff U, Stoylen A, Loennechen JP et al. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation 2007; 115: 3086-3094.

Wonisch M, Hofmann P, Fruhwald FM et al. Influence of beta-blocker use on percentage of target heart rate exercise prescription. Eur J Cardiovasc Prev Rehabil 2003; 10: 296-301.

ELIGIBILITY:
Inclusion Criteria:

* Veteran or non-veteran;
* Presence of all 3 cardinal features of Parkinson's disease (resting tremor, bradykinesia, and rigidity), which have to be asymmetrical;
* Hoehn and Yahr Scale stage I-III;
* Men or women aged 50-80 capable of performing the planned exercise programs;
* Intention to remain in the local area over the study period;
* Stable dopaminergic treatment regimen for at least 4 weeks prior to baseline without any clinical need for medication adjustment at the time of screening

Exclusion Criteria:

* Secondary parkinsonism;
* Parkinson-plus syndromes;
* MMSE score <24;
* Participating in a aerobic exercise program;
* An unstable dosage of drugs active in the central nervous system (e.g., anxiolytics, antidepressants) during the 60 days before the baseline visit;
* Participation in drug studies or the use of investigational drugs within 30 days before screening; structural brain disease;
* Active epilepsy;
* Acute illness or active, confounding medical, neurological, or musculoskeletal conditions; alcoholism or other forms of drug addiction;
* Inability to complete the graded exercise test;
* Lack of medical clearance from our pulmonologist;
* Intention to move or take a >1 month vacation during the study period;
* Contraindications to MRI or claustrophobia requiring sedation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ergun Y. Uc, MD, Principal Investigator — VA Medical Center, Iowa City
Locations (1):
- VA Medical Center, Iowa City, Iowa City, Iowa, United States

REFERENCES:
- [Result] Uc EY, Doerschug KC, Magnotta V, Dawson JD, Thomsen TR, Kline JN, Rizzo M, Newman SR, Mehta S, Grabowski TJ, Bruss J, Blanchette DR, Anderson SW, Voss MW, Kramer AF, Darling WG. Phase I/II randomized trial of aerobic exercise in Parkinson disease in a community setting. Neurology. 2014 Jul 29;83(5):413-25. doi: 10.1212/WNL.0000000000000644. Epub 2014 Jul 2. PMID 24991037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After phone screening, we evaluated 104 eligible candidates in-person (90 community responders to newspaper advertisements and 14 clinic patients).
Pre-assignment Details: Of the 104 consented candidates, 60 participants started the intervention. Thirty-six candidates did not meet eligibility criteria and 8 declined participation due to time commitment.
Groups:
- Continuous Training - Years 1 & 2: The duration of exercise sessions (3x/week) was advanced from 15 to 45 minutes over the first 6 weeks. Participants were asked to wear electronic heart rate and walking speed monitors (Polar RS400, Kempele, Finland) and fill out diaries for each session. The goal for continuous training was to remain within 70-80% of HRmax throughout the session.
- Interval Training - Years 1 & 2: The duration of exercise sessions (3x/week) was advanced from 15 to 45 minutes over the first 6 weeks. Participants were asked to wear electronic heart rate and walking speed monitors (Polar RS400, Kempele, Finland) and fill out diaries for each session. Interval trainees alternated every 3 minutes between slower (60-70% of HRmax) and faster (80-90% of HRmax) walking.
- Continuous Training - Year 3: Participant were assigned to continuous training without randomization.
Period: Years 1 & 2
Arm/Group | Continuous Training - Years 1 & 2 | Interval Training - Years 1 & 2 | Continuous Training - Year 3
Started | 21 | 22 | 0
Completed | 18 | 17 | 0
Not Completed | 3 | 5 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0
Not completed — Adverse Event | 0 | 3 | 0
Period: Year 3
Arm/Group | Continuous Training - Years 1 & 2 | Interval Training - Years 1 & 2 | Continuous Training - Year 3
Started | 0 | 0 | 17
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of subjects.
Groups:
- Continuous Training-Years 1 & 2: Participants who were randomized to continuous training in the first 2 years of the study.
- Interval Training -Years 1 & 2: Participants who were randomized to interval training in the first 2 years of the study.
- Continuous-Year 3: Participants who were assigned to continuous training in the third year of the study without randomization. Due to potentially increased risk of knee pain without additional fitness benefits, we dropped the interval group for the third year.
- Total: Total of all reporting groups
Arm/Group | Continuous Training-Years 1 & 2 | Interval Training -Years 1 & 2 | Continuous-Year 3 | Total
Number analyzed (Participants) | 21 | 22 | 17 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (7.5) | 64.7 (5.2) | 63.7 (4.9) | 65.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 6 | 19
  Male | 15 | 15 | 11 | 41
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 17 | 60
Education [Mean (Standard Deviation); unit: years] | 15.9 (2.3) | 14.6 (2.3) | 14.8 (2.1) | 15.1 (2.3)
Disease duration (years) [Mean (Standard Deviation); unit: years] | 8.0 (6.3) | 5.3 (3.5) | 2.8 (2.5) | 5.5 (4.9)
modified Hoehn-Yahr Scale [Median (Full Range); unit: units on a scale] — Modified Hoehn and Yahr Scale (higher values are worse) 1.0: Unilateral involvement only 1.5: Unilateral and axial involvement 2.0: Bilateral involvement without impairment of balance 2.5: Mild bilateral disease with recovery on pull test 3.0: Mild to moderate bilateral disease; some postural instability; physically independent 4.0: Severe disability; still able to walk or stand unassisted 5.0: Wheelchair bound or bedridden unless aided
  units on a scale | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.5] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
UPDRS- Section III score [Mean (Standard Deviation); unit: units on a scale] — Unified Parkinson's Disease Rating Scale (UPDRS) is an ordinal scale with all items scored from 0=normal function to 4=very severely disabled. Section III: UPDRS motor section is based on physical examination evaluates the components of parkinsonism (tremor, rigidity, bradykinesia, gait/posture). There are 27 items resulting in a maximum score of 108 (range 0-108). Higher scores are worse.
  units on a scale | 19.6 (9.9) | 18.9 (10.5) | 17.0 (10.0) | 18.6 (10.0)
Levodopa equivalent/day [Mean (Standard Deviation); unit: mg/day] — Total antiparkinsonian treatment daily dose expressed in levodopa equivalents per Tomlinson et al (PMID:21069833)
  mg/day | 531 (383) | 601 (273) | 394 (334) | 540 (380)
VO2max [Mean (Standard Deviation); unit: ml/min/kg] | 23.4 (5.6) | 25.1 (8.2) | 27.8 (3.7) | 25.2 (6.5)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — Score ranges from 0-30. Higher scores are better.
  units on a scale | 24.7 (2.8) | 24.2 (3.0) | 24.5 (2.9) | 24.5 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Aerobic Fitness
Description: VO2max after the training - VO2max at baseline (Adjusted for levodopa-equivalent, year, training mode, setting).
  Please see publication PMID: 24991037 for details.
Time Frame: 6 months
Population: Because all treatment arms were designed to deliver a similar average aerobic intensity, we planned to pool a priori all completers from the Continuous and Interval Training Arms for all analyses.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Groups:
- Completers: The participants who completed 6 months of aerobic training
Arm/Group | Completers
Number analyzed (Participants) | 49
ml/min/kg | 1.56 (2.74)
Statistical Analysis 1: Comparison: Completers; Sample size was estimated using 80% power to detect an effect size of 0.66 SD in VO2max (estimated improvement=10% /estimated SD of change=15%) within each arm at alpha=0.05 and an attrition rate of 25%; Test type: Superiority or Other; p < 0.001, Regression, Linear — Because all treatment arms were designed to deliver a similar average aerobic intensity, we planned to pool a priori all completers from the Continuous and Interval Training Arms for analysis

2. Secondary Outcome: Change in 7 Meter Walk Time
Description: Time complete the 7 m Walk test after 6 months aerobic training - Time complete the 7 m Walk test at baseline
Time Frame: 6 months
Population: See PMID: 24991037
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Completers: The participants who completed 6 months of aerobic training. Because all treatment arms were designed to deliver a similar average aerobic intensity, we planned to pool a priori all completers from the Continuous and Interval Training Arms for analysis.
Arm/Group | Completers
Number analyzed (Participants) | 49
seconds | -0.85 (0.94)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p < 0.001, Regression, Linear

3. Secondary Outcome: Change in the UPDRS Section I Score
Description: =Score after 6 months training - baseline score Unified Parkinson's Disease Rating Scale (UPDRS) is an ordinal scale with all items scored from 0=normal function to 4=very severely disabled. It has 3 sections: I) Mental, Behavior, and Mood: Comprises four questions on intellectual impairment, thought disorder, depression, and apathy (scores range 0-16). II) The Activities of Daily Living (ADL) subscale is based on interview and comprises 13 items (scores range 0-52). III) UPDRS motor section is based on physical examination evaluates the components of parkinsonism (tremor, rigidity, bradykinesia, gait/posture). There are 27 items resulting in a maximum score of 108. Higher scores are worse.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | -0.5 (1.6)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.029, Regression, Linear

4. Secondary Outcome: Change in UPDRS Section II Score
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | -0.4 (2.4)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.271, Regression, Linear

5. Other Pre Specified Outcome: Change in Fatigue Severity Scale Score
Description: =Score after 6 months of training - baseline score. The Fatigue Severity Scale (FSS) is a self-administered unidimensional generic 9-item fatigue rating scale. These are rated on a seven-grade Likert scale of which only the respective ends are defined (''completely disagree''=1 to ''completely agree''=7). The total FSS score represents the mean score of each of the nine items, yielding a score range between 1 and 7, higher scores indicating a higher level of fatigue.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | -0.29 (1.29)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.070, Regression, Linear — unadjusted p-value=0.009

6. Other Pre Specified Outcome: Change in Geriatric Depression Scale Score
Description: =Score after 6 months training - score at baseline. The Geriatric Depression Scale (GDS)-short form is a 15 item yes/no questionnaire. The range is 0-15 and scores >5 suggest depression. Higher scores are worse.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | -2.09 (2.33)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p < 0.001, Regression, Linear

7. Other Pre Specified Outcome: Change in Parkinson's Disease Quality of Life Scale (PDQUALIF) Score
Description: = PDQUALIF score after 6 months training - baseline score The PDQUALIF is a 32 item questionnaire resulting in 7 factors. . Subjects rate themselves between 1 (most favorable) and 5 (least favorable) on a Likert scale. Factor scores are standardized to100 and lower scores are better. The outcome measure is the average of these 7 factor scores.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | -1.62 (3.95)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.006, Regression, Linear

8. Secondary Outcome: Change in the UPDRS Section III Score
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | -3.4 (7.0)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.002, Regression, Linear

9. Secondary Outcome: Change in the Total UPDRS Score
Description: =Score after 6 months training - baseline score The total UPDRS score is calculated by adding Section I, Section II, and Section III scores (below). Higher scores are worse. The score ranges 0-176.
  Unified Parkinson's Disease Rating Scale (UPDRS) is an ordinal scale with all items scored from 0=normal function to 4=very severely disabled. It has 3 sections: I) Mental, Behavior, and Mood: Comprises four questions on intellectual impairment, thought disorder, depression, and apathy (scores range 0-16). II) The Activities of Daily Living (ADL) subscale is based on interview and comprises 13 items (scores range 0-52). III) UPDRS motor section is based on physical examination evaluates the components of parkinsonism (tremor, rigidity, bradykinesia, gait/posture). There are 27 items resulting in a maximum score of 108.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | -3.8 (7.4)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.003, Regression, Linear; Adjusted for change in total daily equivalent levodopa dose

10. Secondary Outcome: Change in the MOCA Score
Description: =Score after 6 months training - baseline score. MOCA=Montreal Cognitive Training Assessment Scores range 0-30, higher is better.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Completers
Number analyzed (Participants) | 49
units on a scale | 0.4 (1.8)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.146, t-test, 2 sided

11. Secondary Outcome: Change in Percent Increase Score (PIS) on Eriksen's Flanker Task
Description: performance on the Eriksen's flanker task (see PMID: 24991037). Participants were asked to identify the orientation of a central arrow cue ('<' or '>'), which was flanked on both sides by two arrow cues that either pointed in the same direction (congruent: <<<<<) or a different direction (incongruent: >><>>). Using reaction times (RT) during congruent and incongruent trials, the PIS was calculated as =((RT_incongruent - RT_congruent) / RT_congruent) * 100. Higher PIS is worse.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage of Increase score
Arm/Group | Completers
Number analyzed (Participants) | 49
Percentage of Increase score | -2.41 (7.26)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.037, Regression, Linear

12. Other Pre Specified Outcome: Change in LEDD (Levodopa Equivalent Daily Dose)
Description: =amount after 6 months training - amount at baseline Total antiparkinsonian treatment daily dose expressed in levodopa equivalents per Tomlinson et al (PMID:21069833). Higher scores are worse.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Completers
Number analyzed (Participants) | 49
mg/day | 34 (114)
Statistical Analysis 1: Comparison: Completers; Test type: Superiority or Other; p = 0.057, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Continuous Training: This group consists of 21 subjects who were randomized to continuous training in the first two years of the study and 17 subjects who were assigned to continuous training without randomization in the third year of the study. Thus, total group size is 38.
- Interval Training: This group consists of 22 subjects who were randomized to interval training in the first two years of the study. No subjects were assigned to the interval training in the third year of the study.
Arm/Group | Continuous Training | Interval Training
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/22
Other Adverse Events (participants affected / at risk) | 1/38 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Training (N=38) | Interval Training (N=22)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) — knee or hip pain. Resolved with rest and analgesics

LIMITATIONS AND CAVEATS:
We adapted our design in response to recruitment challenges and preliminary results over the course of the study. This uncontrolled study cannot prove efficacy, but provides guidance for a future Phase III study on aerobic exercise in PD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No